CLINICAL TRIAL: NCT03642743
Title: Patient Satisfaction With Two and Six Week Postoperative Follow up Appointments After Benign Minimally Invasive Hysterectomy Versus Two Week Postoperative Visit Alone: a Randomized Controlled Trial
Brief Title: Patient Satisfaction With Postoperative Follow up After Minimally Invasive Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Shan Biscette, Associate Professor of Gynecology, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18.0481
Record Dates: First submitted 2018-05-02; First posted 2018-08-22 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Minimally Invasive Surgery; Hysterectomy; Postoperative; Satisfaction
Keywords: hysterectomy; minimally invasive surgery; gynecology; satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two and six week follow up (Experimental): Patients will be assigned to routine two and six week postoperative follow up appointments
  Interventions: Other: postoperative follow up appointment
- Six week follow up only (Experimental): Patients will be assigned to a single six week postoperative follow up appointment
  Interventions: Other: postoperative follow up appointment

INTERVENTIONS:
Other: postoperative follow up appointment — Comparison of two and six week postoperative follow up versus a six week postoperative follow up alone

SUMMARY:
This prospective, randomized control trial will evaluate patient satisfaction with the number of postoperative follow up visits after minimally invasive hysterectomy for the treatment of non-cancerous conditions at an urban academic hospital in Louisville, Kentucky. Patients will be randomized to receive either a two and six week postoperative follow up visits versus a postoperative follow up visit at six weeks alone.

DETAILED DESCRIPTION:
The objective of follow up appointments following benign gynecologic surgery is to ensure adequate postoperative recovery, assess additional patient concerns, and to identify and manage any delayed postoperative complications. There is limited literature addressing short-term postoperative follow up for benign gynecologic surgery, particularly those performed through a minimally invasive approach.

The benefits of minimally invasive surgery includes shorter operative time, reduced hospital stay, improved cosmesis, and faster recovery especially when combined with enhanced recovery after surgery (ERAS) protocols. However, this does not negate the need for follow up. Although no consensus exists on the appropriate frequency and number of postoperative appointments, there is no debate on its value.

Due to lack of evidence on this issue, the number and frequency of postoperative appointments is currently dependent on surgeon preference, type of procedure performed and complications encountered intraoperatively and postoperatively, which could lead to patient confusion and unnecessary cost and hassle.

For this reason, investigation of outcomes based on the number and frequency of postoperative follow up visits may improve optimal patient satisfaction, improve compliance and provide early detection of postoperative complications. Such knowledge could serve to mitigate efforts to develop and implement protocols to improve compliance with postoperative follow-up care, potentially reduce emergency room visits, readmissions, empower patients and reduce cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients of University of Louisville gynecology providers age 18-70 who are planning to undergo a minimally invasive hysterectomy for benign indications.
* Incident surgery must be performed at the University of Louisville Hospital (or affiliated hospital attended by a provider affiliated with the academic department).

Exclusion Criteria:

* Patients with decreased mental capacity who are unable to consent.
* Patients who do not have sufficient English proficiency to complete or understand informed consent for the surgery or study questionnaires.
* Patients with unreliable access to a telephone.
* Patients with significant medical comorbidities that would necessitate more frequent follow up.
* Patients for whom the planned number of follow ups have been pre-determined at the pre-operative visit due to a certain medical need or condition.
* Patients who report an inability to comply with postoperative follow up in either group to which they could be randomized.
* Women who decide at their preoperative visit they do not desire or cannot undergo benign gynecologic surgery as scheduled.
* Women who have medical contraindication to undergoing the benign gynecologic surgery that was planned prior, as determined in their best interest by their provider

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 6 weeks
  To assess patient satisfaction with the number of postoperative follow up office visits after minimally invasive hysterectomy for benign indications utilizing the Surgical Care - Consumer Assessment of Healthcare Providers and Systems (CAHPS) Clinician & Group Survey.

SECONDARY OUTCOMES:
Postoperative complication rate | 6 weeks
  Determine the type and number of postoperative complications as assessed using the Clavien-Dindo Classification system has been selected as a validated and objective measure to collect data pertaining to postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Shan Biscette, MD, Principal Investigator — University of Louisville School of Medicine
Locations (1):
- Health Care Outpatient Center and University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu JM, Wechter ME, Geller EJ, Nguyen TV, Visco AG. Hysterectomy rates in the United States, 2003. Obstet Gynecol. 2007 Nov;110(5):1091-5. doi: 10.1097/01.AOG.0000285997.38553.4b. PMID 17978124
- [Result] Cohen SL, Ajao MO, Clark NV, Vitonis AF, Einarsson JI. Outpatient Hysterectomy Volume in the United States. Obstet Gynecol. 2017 Jul;130(1):130-137. doi: 10.1097/AOG.0000000000002103. PMID 28594764
- [Result] Aarts JW, Nieboer TE, Johnson N, Tavender E, Garry R, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2015 Aug 12;2015(8):CD003677. doi: 10.1002/14651858.CD003677.pub5. PMID 26264829
- [Result] Slankamenac K, Graf R, Puhan MA, Clavien PA. Perception of surgical complications among patients, nurses and physicians: a prospective cross-sectional survey. Patient Saf Surg. 2011 Nov 22;5(1):30. doi: 10.1186/1754-9493-5-30. PMID 22107603
- [Result] Bateman AG, Neilens H, Gericke CA, George J, Freeman RM. Is there a need for postoperative follow-up after routine urogynaecological procedures? Patients will self-present if they have problems. Int Urogynecol J. 2014 Mar;25(3):381-6. doi: 10.1007/s00192-013-2229-1. Epub 2013 Oct 9. PMID 24105409
- [Result] Bromage SJ, Napier-Hemy RD, Payne SR, Pearce I. Outpatient follow up appointments; are we using the resources effectively? Postgrad Med J. 2006 Jul;82(969):465-7. doi: 10.1136/pgmj.2005.043547. PMID 16822924
- [Result] McVay MR, Kelley KR, Mathews DL, Jackson RJ, Kokoska ER, Smith SD. Postoperative follow-up: is a phone call enough? J Pediatr Surg. 2008 Jan;43(1):83-6. doi: 10.1016/j.jpedsurg.2007.09.025. PMID 18206461
- [Result] Scott AR, Rush AJ 3rd, Naik AD, Berger DH, Suliburk JW. Surgical follow-up costs disproportionately impact low-income patients. J Surg Res. 2015 Nov;199(1):32-8. doi: 10.1016/j.jss.2015.04.013. Epub 2015 Apr 10. PMID 26013443
- [Result] Tevis SE, Kennedy GD, Kent KC. Is There a Relationship Between Patient Satisfaction and Favorable Surgical Outcomes? Adv Surg. 2015;49(1):221-33. doi: 10.1016/j.yasu.2015.03.006. PMID 26299501
- [Result] Shirley ED, Sanders JO. Patient satisfaction: Implications and predictors of success. J Bone Joint Surg Am. 2013 May 15;95(10):e69. doi: 10.2106/JBJS.L.01048. PMID 23677370
- [Result] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Barrie A, Freeman AH, Lyon L, Garcia C, Conell C, Abbott LH, Littell RD, Powell CB. Classification of Postoperative Complications in Robotic-assisted Compared With Laparoscopic Hysterectomy for Endometrial Cancer. J Minim Invasive Gynecol. 2016 Nov-Dec;23(7):1181-1188. doi: 10.1016/j.jmig.2016.08.832. Epub 2016 Sep 9. PMID 27621195
- [Result] Hernandez Alava M, Wailoo A, Grimm S, Pudney S, Gomes M, Sadique Z, Meads D, O'Dwyer J, Barton G, Irvine L. EQ-5D-5L versus EQ-5D-3L: The Impact on Cost Effectiveness in the United Kingdom. Value Health. 2018 Jan;21(1):49-56. doi: 10.1016/j.jval.2017.09.004. Epub 2017 Oct 18. PMID 29304940
- [Result] Jiang N, Malkin BD. Use of Lean and CAHPS Surgical Care Survey to Improve Patients' Experiences with Surgical Care. Otolaryngol Head Neck Surg. 2016 Nov;155(5):743-747. doi: 10.1177/0194599816657051. Epub 2016 Jun 21. PMID 27329420
- [Result] McCaughey D, Stalley S, Williams E. Examining the effect of EVS spending on HCAHPS scores: a value optimization matrix for expense management. J Healthc Manag. 2013 Sep-Oct;58(5):320-34; discussion 334-5. PMID 24195341
- [Result] Schmocker RK, Cherney Stafford LM, Siy AB, Leverson GE, Winslow ER. Understanding the determinants of patient satisfaction with surgical care using the Consumer Assessment of Healthcare Providers and Systems surgical care survey (S-CAHPS). Surgery. 2015 Dec;158(6):1724-33. doi: 10.1016/j.surg.2015.06.018. Epub 2015 Jul 17. PMID 26195107
- [Result] Sundararajan V, Henderson T, Perry C, Muggivan A, Quan H, Ghali WA. New ICD-10 version of the Charlson comorbidity index predicted in-hospital mortality. J Clin Epidemiol. 2004 Dec;57(12):1288-94. doi: 10.1016/j.jclinepi.2004.03.012. PMID 15617955
- [Result] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Result] Becerra Perez MM, Menear M, Brehaut JC, Legare F. Extent and Predictors of Decision Regret about Health Care Decisions: A Systematic Review. Med Decis Making. 2016 Aug;36(6):777-90. doi: 10.1177/0272989X16636113. Epub 2016 Mar 14. PMID 26975351
- [Result] Agdi M, Al-Ghafri W, Antolin R, Arrington J, O'Kelley K, Thomson AJ, Tulandi T. Vaginal vault dehiscence after hysterectomy. J Minim Invasive Gynecol. 2009 May-Jun;16(3):313-7. doi: 10.1016/j.jmig.2009.01.006. Epub 2009 Mar 14. PMID 19285921
- [Result] AAGL Advancing Minimally Invasive Gynecology Worldwide. AAGL position statement: route of hysterectomy to treat benign uterine disease. J Minim Invasive Gynecol. 2011 Jan-Feb;18(1):1-3. doi: 10.1016/j.jmig.2010.10.001. Epub 2010 Nov 6. No abstract available. PMID 21059487
- [Result] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801